CLINICAL TRIAL: NCT04109898
Title: Comparison of Ease of I-gel Insertion With Two Different Techniques in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dileep Kumar, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-1878-4900.
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Airway Morbidity
Keywords: airway management; I-gel; anaesthesia
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard I-gel insertion technique (No Intervention): Investigator will apply the recommended (standard) I-gel insertion technique in patients
- Modified I-gel insertion technique (Experimental): Investigator will apply the modified (interventional) I-gel insertion technique in patients
  Interventions: Device: Supraglottic airway device (I-gel) insertion

INTERVENTIONS:
Device: Supraglottic airway device (I-gel) insertion — Modified I-gel insertion technique believed to be easier and non traumatic in anaesthetised patients.
  Arms: Modified I-gel insertion technique

SUMMARY:
Study will evaluate the I-gel airway device standard insertion technique versus interventional (modified jaw thurst) insertion technique in adult patients. The half of the patients will receive standard and other half will receive the modified jaw thrust insertion technique

DETAILED DESCRIPTION:
The I-gel is used to provide the oxygenation and ventilation in anaesthetised patients. The inventor suggested insertion technique is called standard technique.

Standard I-gel insertion technique: I-gel insertion will be performed by firmly grasping the lubricated I-gel along the integral bite block site. I-gel cuff outlet will face towards the patient's chin and before insertion chin will be gently pressed down. The I-gel soft tip will be introduced into patient's mouth in a direction towards the hard palate. Then I-gel will be slide downwards and backwards along the hard palate with a continuous but gentle push until a definitive resistance is felt.

Modified jaw thrust technique: I-gel insertion will be performed by firmly grasping the lubricated I-gel along the integral bite block. I-gel cuff outlet will face towards the patient's chin and before insertion chin will be gently pressed down. The I-gel soft tip will be introduced into patient's mouth in a direction towards the hard palate and it slides gently into the oropharynx. I-gel will be left in oral cavity and both hands will be used to thrust the jaw by lifting the angle of mandible with little fingers and other fingers to stabilize the jaw then both thumbs will used to apply the balance force towards the final I-gel placement position by looking at the integral bite block mark at incisor teeth level.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients.
* Age 16 years to 60 years.
* Patient scheduled for elective surgical procedure.

Exclusion Criteria:

* Gastroesophageal reflux disorders
* Obesity BMI more than 30.
* Pregnancy
* Reactive airway disease/asthma
* Patients with mallampati score III & IV
* Anticipated difficult airway
* Emergent surgery.
* Known allergic to isoflurane and propofol.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2019-09-07 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
adverse airway events | 5 minutes
  All study patients will be monitored for I-gel insertion resistance, insertion time duration, insertion attempts.

SECONDARY OUTCOMES:
adverse airway events | 60 minutes
  All study patients will be monitored forI-gel insertion complications such as an laryngospasm, hypoxemia (Sp02<92%) and trauma to surrounding airway structures will be observe as blood stained I-gel at removal.

CONTACTS AND LOCATIONS:
Overall Officials: dileep kumar, MD, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan